CLINICAL TRIAL: NCT01383005
Title: Treatment Perception of QD Dosed Kaletra (Tablets) Based Treatment in HIV Infected Patients. Observational Cross-Sectional Study (QD-KAPITAL)
Brief Title: Treatment Perception of QD (Once a Day) Dosed Kaletra (Tablets)
Acronym: QD-Kapital
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Triaca Magna, SA (Unknown)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-752
Record Dates: First submitted 2011-05-31; First posted 2011-06-28 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-04

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: Treatment satisfaction; Adherence to treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Kaletra (LPV/r) QD as First Kaletra Treatment: HIV-infected participants treated with lopinavir/ritonavir once daily (LPV/r QD) from ≥3 months to <2 years who had not been treated with any of the following: LPV/r twice daily (BID), a protease inhibitor, or a ritonavir-boosted protease inhibitor.
- Kaletra (LPV/r) QD from Kaletra BID: HIV-infected participants treated with LPV/r from ≥3 months to <2 years who had initiated on LPV/r BID and at any time within this period (but at least 3 months before inclusion in the study) had changed dosing from BID to QD.

SUMMARY:
Both twice-a-day (BID) and once-a-day (QD) dosing are approved in Europe for the protease inhibitor lopinavir/ritonavir (LPV/r; Kaletra®).

Since once-a-day dosing is actually a driver for human immunodeficiency virus (HIV)-infected patients to request a specific antiretroviral, the aim of this study is to assess both patient's perception of and adherence to Kaletra once-a-day, as well as with which factors they are related.

DETAILED DESCRIPTION:
This is a multicenter, post-marketing, observational, cross-sectional (single visit) study in HIV-infected patients treated with a combination of antiretroviral treatment (ART) containing LPV/r 200/50 mg tablets dosed QD for at least 12 weeks to assess the participants' satisfaction and adherence level with LPV/r QD ART as measured by specific validated participant questionnaires.

As this is a non-interventional study, the decision to enroll a participant was separate from the decision to treat the subject with LPV/r. Prescription of LPV/r and duration of treatment were the responsibility of the treating physician.

In addition, the overall study population was compared to Cohort 2 (394 patients on LPV/r BID for ≥3 months to <2 years) from KAPITAL2, a post-marketing observational, cross-sectional, single visit, multicenter, national study. For further details on this study, please see: Casado JL, Griffa L, Cabrero E, Burgos A, Norton M and the KAPITAL 2 Collaborative Group. A study of treatment satisfaction reported by patients on lopinavir/r anchored regimens and physicians who provide HIV care (KAPITAL 2). 9th International Congress on Drug Therapy in HIV Infection. 9th International Congress on Drug Therapy in HIV Infection. Glasgow, 2008.#P080.

ELIGIBILITY:
Inclusion criteria:

1. Men or women aged 18 years or older, HIV-infected.
2. Patients who were under LPV/r Highly Active Anti-Retroviral Therapy (HAART) for 3 to 24 months before study visit:

   Cohort 1: patients on LPV/r QD since they started the LPV/r regimen and who were naïve to protease inhibitor (PI) therapy.* Cohort 2: patients who previously started on LPV/r BID (maximum of 24 months before study) and switched to LPV/r QD (at least 3 months before the study visit).*
3. Patients who were able to complete questionnaires by themselves.
4. Patients who signed/dated informed consent to participate in the study.

   * NOTE: Patients who were taking LPV/r QD should have had no more than 3 protease inhibitor mutations by the time the treatment with this LPV/r dosing was initiated.

Exclusion criteria:

1. Patients who were on LPV/r monotherapy or bi-therapy or on BID dosing at time of study visit.
2. Patients who were using another LPV/r formulation different from 200/50 LPV/r mg tablets.
3. Patients who were participating in any other clinical trial or postmarketing observational study (PMOS).
4. Patients who were unable to read and/or write.
5. Patients who were under treatment interruption. Patients who have stopped LPV-therapy for more than 3 months in the 12 months preceding study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients regularly visiting Spanish hospital/clinic physicians and treated with lopinavir/ritonavir once-a-day regimens.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Burgos, PhD, Study Director — AbbVie S.L.U.
Locations (20):
- Spain (20):
  - Site Ref # / Investigator 52274, A Coruña
  - Site Ref # / Investigator 52363, Barakaldo
  - Site Ref # / Investigator 52271, Barcelona
  - Site Ref # / Investigator 52270, Barcelona
  - Site Ref # / Investigator 52362, Cartagena
  - Site Ref # / Investigator 53650, Castellon
  - Site Ref # / Investigator 52273, Ferrol (A Coruna)
  - Site Ref # / Investigator 52264, Granada
  - Site Ref # / Investigator 52262, Jaén
  - Site Ref # / Investigator 52263, Jerez de La Frontera (Cadiz)
  - Site Ref # / Investigator 52267, L'Hospitalet de Llobregat
  - Site Ref # / Investigator 52345, Madrid
  - Site Ref # / Investigator 52275, Madrid
  - Site Ref # / Investigator 52302, Madrid
  - Site Ref # / Investigator 52343, Madrid
  - Site Ref # / Investigator 52344, Madrid
  - Site Ref # / Investigator 53648, Murcia
  - Site Ref # / Investigator 52268, Reus (Tarragona)
  - Site Ref # / Investigator 52272, Valencia
  - Site Ref # / Investigator 52266, Zaragoza

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 97 participants were enrolled; 3 participants who did not meet the inclusion criteria for treatment duration were excluded.
Period: Overall Study
Arm/Group | Kaletra (LPV/r) QD as First Kaletra Treatment | Kaletra (LPV/r) QD From Kaletra BID
Started | 34 | 60
Completed | 34 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kaletra (LPV/r) QD as First Kaletra Treatment | Kaletra (LPV/r) QD From Kaletra BID | Total
Number analyzed (Participants) | 34 | 60 | 94
Age Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.4) | 39.9 (8.8) | 38.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 21 | 30
  Male | 25 | 39 | 64

OUTCOME MEASURES:

1. Primary Outcome: Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Individual Item Scores for the Overall Study Population
Description: Participant treatment satisfaction was measured using the HIVTSQ, which consists of 10 items (1-Satisfaction, 2-HIV Control, 3-Adverse Effects, 4-Level of Demand, 5-Convenience, 6-Flexibility, 7-Knowledge, 8-Life Habits, 9-Recommendability, and 10-Willingness to Continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). Each single item was considered for the evaluation of the primary outcome.
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants with complete data. n=number of participants with complete data for given HIVTSQ item.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Overall Study Population: HIV-infected participants treated with lopinavir/ritonavir once daily (LPV/r QD) from ≥3 months to <2 years who had not been treated with any of the following: LPV/r twice daily (BID), a protease inhibitor, or a ritonavir-boosted protease inhibitor.
  Also, HIV-infected participants treated with LPV/r from ≥3 months to <2 years who had initiated on LPV/r BID and at any time within this period (but at least 3 months before inclusion in the study) had changed dosing from BID to QD.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 94
units on a scale
  Item 1: Satisfied (n=93) | 5.0 (1.2)
  Item 2: HIV Control (n=93) | 5.4 (1.0)
  Item 3: Adverse Effects (n=93) | 4.8 (1.3)
  Item 4: Demanding (n=94) | 2.4 (2.3)
  Item 5: Convenient (n=94) | 4.8 (1.4)
  Item 6: Flexible (n=94) | 4.2 (1.9)
  Item 7: Knowledge (n=93) | 4.6 (1.4)
  Item 8: Life Habits (n=94) | 4.9 (1.3)
  Item 9: Would Recommend (n=94) | 5.1 (1.2)
  Item 10: Willing to Continue (n=94) | 5.0 (1.5)

2. Secondary Outcome: Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Individual Item Scores Comparison Between Cohorts
Description: The HIVTSQ consists of 10 items (1-Satisfaction, 2-HIV Control, 3-Adverse Effects, 4-Level of Demand, 5-Convenience, 6-Flexibility, 7-Knowledge, 8-Life Habits, 9-Recommendability, and 10-Willingness to Continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). The mean score per item was compared between cohorts.
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants with complete data. n=number of participants with complete data for given HIVTSQ item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kaletra (LPV/r) QD as First Kaletra Treatment | Kaletra (LPV/r) QD From Kaletra BID
Number analyzed (Participants) | 34 | 60
units on a scale
  Item 1: Satisfied (n=33, 60) | 5.0 (27.7) | 5.1 (18.3)
  Item 2: HIV Control (n=33, 60) | 5.4 (18.1) | 5.5 (16.1)
  Item 3: Adverse Effects (n=33, 60) | 4.8 (24.0) | 5.1 (19.6)
  Item 4: Demanding (n=34, 60) | 2.4 (38.4) | 2.5 (38.3)
  Item 5: Convenient (n=34, 60) | 4.8 (24.0) | 5.0 (21.6)
  Item 6: Flexible (n=34, 60) | 4.2 (32.5) | 4.3 (30.6)
  Item 7: Knowledge (n=33, 60) | 4.6 (23.6) | 4.7 (22.1)
  Item 8: Life Habits (n=34, 60) | 4.9 (22.9) | 5.0 (21.6)
  Item 9: Would Recommend (n=34, 60) | 5.1 (21.4) | 5.3 (19.7)
  Item 10: Willing to Continue (n=34, 60) | 5.0 (26.4) | 5.1 (23.5)

3. Primary Outcome: Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ)Dimension (Overall Satisfaction, General/Clinical Satisfaction, Lifestyle) Scores for the Overall Study Population
Description: The HIVTSQ consists of 10 items (1-Satisfaction, 2-HIV Control, 3-Adverse Effects, 4-Level of Demand, 5-Convenience, 6-Flexibility, 7-Knowledge, 8-Life Habits, 9-Recommendability, and 10-Willingness to Continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). The items are aggregated to 3 different dimensions: the Overall Satisfaction dimension, with a maximum score of 54 (items 1, 2, 3, 5, 6, 7, 8, 9 and 10); General/Clinical Satisfaction dimension, with a maximum score of 30 (items 1, 2, 3, 9 and 10); Lifestyle dimension, with a maximum score of 24 (items 5, 6, 7 and 8). Each dimension was considered for the evaluation of the primary outcome. For each participant, each dimension score was calculated as a sum of the individual item scores.
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants with complete data. n=number of participants with complete data for given HIVTSQ item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Population
Number analyzed (Participants) | 93
units on a scale
  Score for Overall Satisfaction (n=92) | 44.4 (7.6)
  Score for General/Clinical Satisfaction (n=93) | 25.5 (4.9)
  Score of Lifestyle (n=93) | 18.6 (4.1)

4. Secondary Outcome: Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Dimension (Overall Satisfaction, General/Clinical Satisfaction, Lifestyle) Scores Comparison Between Cohorts
Description: The HIVTSQ consists of 10 items (1-Satisfaction, 2-HIV Control, 3-Adverse Effects, 4-Level of Demand, 5-Convenience, 6-Flexibility, 7-Knowledge, 8-Life Habits, 9-Recommendability, and 10-Willingness to Continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). The items are aggregated to 3 different dimensions: the Overall Satisfaction dimension, with a maximum score of 54 (items 1, 2, 3, 5, 6, 7, 8, 9 and 10); General/Clinical Satisfaction dimension, with a maximum score of 30 (items 1, 2, 3, 9 and 10); Lifestyle dimension, with a maximum score of 24 (items 5, 6, 7 and 8). The mean score per dimension was compared between cohorts.
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants with complete data. n=number of participants with complete data for given HIVTSQ item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kaletra (LPV/r) QD as First Kaletra Treatment | Kaletra (LPV/r) QD From Kaletra BID
Number analyzed (Participants) | 33 | 60
units on a scale
  Score for Overall Satisfaction (n=32, 60) | 43.3 (7.9) | 45.0 (7.5)
  Score for General/Clinical Satisfaction (n=33, 60) | 24.4 (5.7) | 26.1 (4.4)
  Score for Lifestyle (n=33, 60) | 18.2 (4.4) | 18.9 (3.9)

5. Secondary Outcome: Number of Days Without Medication, Per Simplified Medication Adherence Questionnaire (SMAQ)
Description: Number of days without medication was assessed by 1 of the 6 items on the patient questionnaire Simplified Medication Adherence Questionnaire (SMAQ): How many full days have you missed your medication since your last visit? (Please see Outcome Measure 6 for details regarding the remaining 5 items on the SMAQ.)
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants with complete data.
Measure: Number; unit: participants
Arm/Group | Kaletra (LPV/r) QD as First Kaletra Treatment | Kaletra (LPV/r) QD From Kaletra BID
Number analyzed (Participants) | 34 | 59
participants
  None | 30 | 36
  One Day | 3 | 8
  More than One Day | 1 | 15

6. Secondary Outcome: Adherence Classification of Participants Per Simplified Medication Adherence Questionnaire (SMAQ)
Description: Participants' adherence was classified according to answers for 5 of 6 items on the participant questionnaire Simplified Medication Adherence Questionnaire (SMAQ): 4 yes/no questions: Do you ever forget to take your medicines? Do you take your medicines at the instructed time? If you ever feel ill, do you stop taking the medication? Have you ever missed your medication during weekends?; plus the following: In the past week, how many times have you missed your medication? (0, 1-2, 3-5, 6-10, >10). (Please see Outcome Measure 5 for details regarding the 6th item on the SMAQ.) Perfect adherence = no dose was forgotten, medication was not skipped for any reason, and the schedule was not modified; adequate adherence = no dose was forgotten, but at least one dose was not taken at the indicated time; poor adherence = one or more doses were not taken.
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants with complete data.
Measure: Number; unit: participants
Arm/Group | Kaletra (LPV/r) QD as First Kaletra Treatment | Kaletra (LPV/r) QD From Kaletra BID
Number analyzed (Participants) | 34 | 60
participants
  Perfect Adherence | 19 | 28
  Adequate Adherence | 11 | 11
  Poor Adherence | 4 | 21

7. Secondary Outcome: Reasons for Starting or Switching to a Lopinavir/Ritonavir Once Daily (LPV/r QD)Regimen
Description: Participants' cumulative reasons for starting or switching to a LPV/r QD regimen were tabulated via the following yes/no questions entered on the case report form by the physician: simplification (simp) as reason to change to LPV/r QD; preference (pref) of patient as reason to change to LPV/r QD; adjustment to other antiretrovirals (adjust to ARV) as reason to change to LPV/r QD; adherence as reason to change to LPV/r QD; patient's lifestyle as reason to change to LPV/r QD; tolerability as reason to change to LPV/r QD.
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants
Measure: Number; unit: participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 94
participants
  Simp+ Pref + Adjust to ARV + Adherence + Lifestyle | 2
  Simp + Pref + Adjust to ARV + Adherence | 3
  Simp + Pref + Adjust to ARV + Lifestyle | 1
  Simp+ Pref + Adherence + Lifestyle | 3
  Simp + Pref + Adherence | 4
  Simp + Pref + Lifestyle | 2
  Simp + Pref | 3
  Simp + Adjust to ARV + Adherence + Lifestyle | 2
  Simp + Adjust to ARV + Adherence | 5
  Simp + Adjust to ARV + Lifestyle | 1
  Simp + Adjust to ARV | 1
  Simp + Adherence + Lifestyle + Tolerability | 1
  Simp + Adherence + Lifestyle | 6
  Simp + Adherence | 12
  Simp + Lifestyle | 1
  Simp + Tolerability | 1
  Simp | 18
  Pref + Adjust to ARV + Adherence + Lifestyle | 1
  Pref + Adjust to ARV | 1
  Pref + Adherence + Lifestyle | 1
  Pref + Adherence | 1
  Pref | 4
  Adjust to ARV + Adherence + Lifestyle | 1
  Adjust to ARV + Lifestyle | 3
  Adjust to ARV | 1
  Adherence + Lifestyle + Tolerability | 1
  Adherence + Lifestyle | 5
  Adherence | 6
  Lifestyle | 3

8. Secondary Outcome: Percentage of Participants With a Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Overall Satisfaction Dimension Mean Score Value of ≥5 and <5
Description: The HIVTSQ consists of 10 items (1-Satisfaction, 2-HIV Control, 3-Adverse Effects, 4-Level of Demand, 5-Convenience, 6-Flexibility, 7-Knowledge, 8-Life Habits, 9-Recommendability, and 10-Willingness to Continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). The items are aggregated to 3 different dimensions. The Overall Satisfaction dimension has a maximum score of 54 (items 1, 2, 3, 5, 6, 7, 8, 9 and 10). The mean of the individual item scores were dichotomized as 'mean score <5 (lower participant perception of LPV/r QD)' and 'mean score ≥5 (high or very high participant perception of LPV/r QD).' The dependent variable of a mean score <5 was correlated with the independent variables of viral load and time on treatment (see Outcome Measures 9 and 10), to determine the factors associated with a participant's lower perception of QD LPV/r treatment.
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 93
percentage of participants
  Mean Score ≥5 | 54.3
  Mean Score <5 | 45.7

9. Secondary Outcome: Viral Load (VL) Change After at Least 12 Weeks of Treatment With the Lopinavir/Ritonavir (LPV/r)
Description: Viral load change was categorized as either 'detectable to undetectable,' 'undetectable to undetectable,' or 'current detectable' (includes participants whose viral load changed from undetectable to detectable and those whose viral load was detectable throughout). This independent variable was correlated with the percentage of participants with the dependent variable of a Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Overall Satisfaction dimension mean score value of <5 (see Outcome Measure 8), to determine the factors associated with a participant's lower perception of QD LPV/r treatment (see statistical analyses for odds ratio).
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants, per responses to the HIVTSQ Overall Satisfaction Dimension
Measure: Number; unit: participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 93
participants
  Detectable to Undetectable | 51
  Undetectable to Undetectable | 16
  Current Detectable | 25
Statistical Analysis 1: Comparison: Overall Study Population; Statistical Analysis 1 presents the risk of a 'mean score <5' on the HIVTSQ overall satisfaction dimension (see Outcome Measure 8) when correlated with a viral load change from 'detectable to undetectable' in the last model of the Wald test; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Degree of freedom is 1 for the independent variable 'viral load change from detectable to undetectable.'; Odds Ratio (OR) = 0.160, 95% CI 2-sided [0.052 to 0.494] — Stepwise procedures forward and backward were used to select variables in the model using entry and exit probabilities of 0.05 and 0.1 respectively. Identical models were obtained by forward and backward selection procedures
Statistical Analysis 2: Comparison: Overall Study Population; Statistical Analysis 2 presents the risk of a 'mean score <5' on the HIVTSQ overall satisfaction dimension (see Outcome Measure 8) when correlated with a viral load change from 'undetectable to undetectable' in the last model of the Wald test; Test type: Superiority or Other; p = 0.072, Regression, Logistic; Degree of freedom is 1 for the independent variable 'viral load change from undetectable to undetectable.'; Odds Ratio (OR) = 0.279, 95% CI 2-sided [0.070 to 1.118] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Mean Number of Days on LPV/r QD
Description: This independent variable was correlated with the percentage of participants with the dependent variable of an HIVTSQ Overall Satisfaction dimension mean score value of <5 (see Outcome Measure 8), to determine the factors associated with a participant's lower perception of QD LPV/r treatment (see statistical analysis for odds ratio).
Time Frame: At the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Population: All participants, per responses to the HIVTSQ Overall Satisfaction Dimension
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Overall Study Population
Number analyzed (Participants) | 92
days | 208.3 (161.2)
Statistical Analysis 1: Comparison: Overall Study Population; Statistical Analysis 1 presents the risk of a 'mean score <5' on the HIVTSQ overall satisfaction dimension (see Outcome Measure 8) when correlated with time on treatment with LPV/r QD in the last model of the Wald test; Test type: Superiority or Other; p = 0.025, Regression, Logistic; Degree of freedom is 1 for the independent variable 'time on LPV/r.'; Odds Ratio (OR) = 0.996, 95% CI 2-sided [0.992 to 0.999] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Comparison of Mean Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Dimension Scores From QD-KAPITAL and KAPITAL2 Studies
Description: Participants' perceptions of the QD and BID LPV/r regimens using data from the overall study population of QD-KAPITAL and from Cohort 2 of a 2007-2008 study, respectively (KAPITAL2, Casado et al. See Detailed Description for full reference). The KAPITAL2 cohort was comprised of HIV-infected participants treated with LPV/r BID from ≥3 months to <2 years for at least 1 month before inclusion in the study. Data for the overall study population of QD-KAPITAL are provided here, but a comparison to Cohort 2 from the KAPITAL2 study is not presented.
Time Frame: at the single study visit, performed after at least 12 weeks of treatment with Kaletra
Population: All participants with evaluable data. n=the number of participants with data for given dimension.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Population
Number analyzed (Participants) | 93
units on a scale
  Overall Satisfaction (n=92) | 44.4 (7.6)
  General/Clinical Satisfaction (n=93) | 25.5 (4.9)
  Lifestyle (n=93) | 18.6 (4.1)

12. Secondary Outcome: Percentage of Participants With Missing Doses During "the Past 4 Days" and "the Last Weekend" in KAPITAL-2 and QD-KAPITAL Studies
Description: Adherence to LPV/r QD therapy (overall study population of QD-KAPITAL) compared with that of LPV/r BID therapy using data of Cohort 2 from a 2007-2008 study, respectively (KAPITAL2, Casado et al. See Detailed Description for full reference). The KAPITAL2 cohort was comprised of HIV-infected participants treated with LPV/r BID from ≥3 months to <2 years for at least 1 month before inclusion in the study. (A full comparison of the adherence between the QD-KAPITAL study and the KAPITAL2 study could not be made due to formal differences in the applied adherence questionnaires; therefore, the above in-common specified item was compared.) Data for the overall study population of QD-KAPITAL are provided here, but a comparison to Cohort 2 from the KAPITAL2 study is not presented.
Time Frame: at the single study visit, performed after at least 12 weeks of treatment with Kaletra
Population: All participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study Population
Number analyzed (Participants) | 94
percentage of participants
  No Missing Doses During Past 4 days | 90.4
  ≥1 Missing Doses During Past 4 days | 9.6
  No Missing Doses During Last Weekend | 90.4
  ≥1 Missing Doses During Last Weekend | 9.6

ADVERSE EVENTS:
Time Frame: Collected at the single study visit, performed after at least 12 weeks of treatment with Kaletra QD
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 13/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study Population (N=94)
Diarrhea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Burning Sensation (General disorders) | 2
Skin Disorders NOS (Skin and subcutaneous tissue disorders) | 1
Sexual Disorder NOS (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.